CLINICAL TRIAL: NCT03645278
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR0532 Tablets in Healthy Subjects
Brief Title: The PK/PD Study of SHR0532 Tablets in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0532-101
Record Dates: First submitted 2018-08-12; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR0532 (Experimental): Up to 5 cohorts of healthy subjects will receive a single dose of oral SHR0532 tablet.
  Interventions: Drug: SHR0532
- Placebo (Experimental): Up to 5 cohorts of healthy subjects will receive a single dose of oral placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0532 — Ascending dose oral adminstration
  Arms: SHR0532
Drug: Placebo — Ascending dose oral administration
  Arms: Placebo

SUMMARY:
In the last four decades, several classes of diuretics have been the first line option for the therapy of widespread hypertension. However, all the classes of diuretics cause alteration of potassium homeostasis. The primary objective of this study is to assess the safety and tolerability of SHR0532 tablets in healthy subjects. In addition, this study will provide information on Pharmacokinetics and Pharmacodynamics of SHR0532 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, aged 18-45
2. subjects have no cardiovascular disease, with sitting blood pressure: 90mmHg ≤SBP<140mmHg and 60mmHg ≤DBP<90mmHg;
3. body mass index (BMI) between 19 to 26, and a total body weight: male ≥50.0 kg and <90.0 kg; female ≥45.0 kg and <90.0 kg
4. Participant in general good health. No clinically significant findings in laboratory parameters or clinically significant abnormality on electrocardiogram, X-ray, Echocardiograph and B-type ultrasonic

Exclusion Criteria:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin > 1.5 x ULN during screening/baseline;
2. Serum creatinine>ULN)during screening/baseline;
3. Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) test positive;
4. Known postural hypotension; the numeric difference of systolic blood pressure between both upper limbs >20mmHg；
5. A clinical history of arrhythmia；subjects with Electrocardiogram QTc prolongation（male>450ms；female>460ms）during screening；
6. A clinical history of hyperuricemia；serum uric acid > the upper limit of normal value (ULN) during screening;
7. A clinical history of diabetes；fasting plasma glucose or hemoglobin A1c exceeded the upper limit of normal value (ULN) during screening;
8. Subjects with previous GI discomfort -abdominal pain, diarrhea, and nausea 3 months prior to screening；
9. A clinical history of acute or chronic kidney disease;
10. Subjects with severe trauma or surgery within 3 months prior to the screening； 11.3 months prior to screening involved in any drug or medical device clinical subjects, or within 5 half-life of drugs (test drug half-life more than 3 months) before screening;

12.Pregnant or Serum β-hCG > 5mIU/mL at baseline or women who are breastfeeding; etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-24 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events | Pre-dose to 5 days after dose administration

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SHR-0532 | Pre-dose to 5 days after dose administration
Maximum observed serum concentration (Cmax) of SHR-0532 | Pre-dose to 5 days after dose administration
Time to maximum observed serum concentration (tmax) of SHR-0532 | Pre-dose to 5 days after dose administration
Time to elimination half-life (t1/2) of SHR-0532 | Pre-dose to 5 days after dose administration
Apparent total clearance of the drug from plasma after oral administration (CL/F) of SHR-0532 | Pre-dose to 5 days after dose administration
Apparent volume of distribution after non-intravenous administration (V/F) of SHR-0532 | Pre-dose to 5 days after dose administration
Renal clearance of the drug from plasma (CLR) of SHR-0532 | Pre-dose to 5 days after dose administration
Cumulative amount of unchanged drug excreted into the urine(Ae) of SHR-0532 | Pre-dose to 5 days after dose administration